CLINICAL TRIAL: NCT00197951
Title: Clinical Trial With Ziprasidone for the Treatment of Psychiatric Pathology, Not Being a Severe Mental Disorder, Associated to Alcohol Dependence Disorder.
Brief Title: Clinical Trial With Ziprasidone for the Treatment of Psychiatric Pathology Associated to Alcoholism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-001056-36
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Depression; Anger; Anxiety; Alcoholism
Keywords: Psychiatric symptoms associated to alcoholism recovery; Alcoholism treatment; Alcohol craving; Relapse to heavy drinking; Abuse of other substances during alcoholism recovery
MeSH Terms: conditions — Depression; Anxiety Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Treatment of psychiatric symptoms associated to alcoholism

SUMMARY:
Alcohol dependent patients show comorbid psychiatric symptoms, related to malfunction of dopamine, norepinephrine and serotonin neurotransmission, during early recovery. Ziprasidone can improve malfunctioning of these disregulated systems, thereby improving anxiety, depression, anhedonia, anger, and alcohol craving.

DETAILED DESCRIPTION:
60 alcohol-dependent patients will be included, once finished alcohol detoxification treatment.Thirty patients will receive ziprasidone treatment, in progressively increasing doses, starting from 40 mg per day, and the other 30 patients will receive placebo, in a double blind procedure

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR criteria for alcohol dependence disorder
* Age between 18 -65 years old.
* Score 7 or higher in the GHQ-28 scale.

Exclusion Criteria:

* More than 30 days without drinking alcohol.
* Severe medical disorders.
* Psychotic or bipolar disorders severely decompensated requiring antipsychotic medication.
* Opiate, cocaine or benzodiazepine dependence disorders, requiring more than one week of detoxification treatment.
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Score opf SCL-90-R psychiatric symptoms scale.

SECONDARY OUTCOMES:
Alcohol consumption (amount and frequency)
Alcohol craving
Other substances consumption

CONTACTS AND LOCATIONS:
Overall Officials: Josep Guardia, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Unidad de Conductas Adictivas//Servicio de Psiquiatría//Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain